CLINICAL TRIAL: NCT01608737
Title: A Phase III, Randomised, Double-blind and Placebo-controlled Study of Once Daily BI 201335 for 12 or 24 Weeks in Combination With Pegylated interferon-a and Ribavirin in Treatment-naive and Prior Relapser Patients With Genotype 1 Chronic Hepatitis C Infection
Brief Title: A Phase III Study of BI201335 in Treatment-naive and Prior Relapser Patients With Chronic Hepatitis C Infection
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 1220.8; 2012-001242-18 (EudraCT Number: EudraCT)
Record Dates: First submitted 2012-05-29; First posted 2012-05-31 (Estimated); Last update posted 2013-02-26 (Estimated); Status verified 2013-02

CONDITIONS: Hepatitis C, Chronic
MeSH Terms: conditions — Hepatitis C, Chronic | interventions — faldaprevir

ARMS (5):
- 2. BI 201335 for 24 weeks (Experimental): BI 201335 once daily low dose for 24 weeks, in combined with PegIFN/RBV for 24 or 48 weeks in treatment-naive patients
  Interventions: Drug: BI 201335
- 3. BI 201335 for 12 weeks (Experimental): BI 201335 once daily high dose for 12 weeks, in combined with PegIFN/RBV for 24 or 48 weeks in treatment-naive patients
  Interventions: Drug: BI 201335
- 1. PegIFN/RBV (Active Comparator): PegIFN/RBV for 48 weeks in treatment-naive patients
  Interventions: Drug: PegIFN/RBV
- 4. PegIFN/RBV (Active Comparator): PegIFN/RBV for 48 weeks in prior relapser patients
  Interventions: Drug: PegIFN/RBV
- 5. BI 201335 for 12 weeks (Experimental): BI 201335 once daily high dose for 12 weeks, in combined with PegIFN/RBV for 24 or 48 weeks in prior relapser patients
  Interventions: Drug: BI 201335

INTERVENTIONS:
Drug: PegIFN/RBV — PegIFN/RBV for 48 weeks
  Arms: 4. PegIFN/RBV
Drug: BI 201335 — BI 201335 once daily high dose for 12 weeks
  Arms: 3. BI 201335 for 12 weeks
Drug: BI 201335 — BI 201335 once daily high dose for 12 weeks
  Arms: 5. BI 201335 for 12 weeks
Drug: PegIFN/RBV — PegIFN/RBV for 48 weeks
  Arms: 1. PegIFN/RBV
Drug: BI 201335 — BI 201335 once daily low dose for 24 weeks
  Arms: 2. BI 201335 for 24 weeks

SUMMARY:
The objectives of this study are:

1. To evaluate the efficacy and safety of two different treatment regimens with BI 201335 (high dose given for 12 weeks or low dose given for 24 weeks both in combination with Pegylated interferon-a and Ribavirin (PegIFN/RBV) as compared to PegIFN/RBV alone in treatment-naïve (TN) chronic genotype 1 hepatitis C virus infected patients.
2. Evaluate the efficacy and the safety of BI 201335 high dose given for 12 weeks in combination with PegIFN/RBV given for 24 to 48 weeks as compared to PegIFN/RBV alone in chronic GT-1 hepatitis C virus infected relapser patients who failed a prior PegIFN/RBV treatment.

ELIGIBILITY:
Inclusion criteria:

1. Chronic hepatitis C infection, diagnosed by positive anti-HCV antibodies and detectable hepatitis C virus (HCV) ribonucleic acid ( RNA) at screening in addition to:

   1. Positive anti-HCV antibodies or detectable HCV RNA at least 6 months prior to screening or,
   2. Liver biopsy consistent with chronic HCV infection
2. HCV genotype 1 infection confirmed by genotypic testing at screening
3. Therapy-naïve to interferon, pegylated interferon, and ribavirin (cohort 1). Or Confirmed prior relapse with an approved dose of PegIFN/RBV(Cohort 2) defined as undetectable HCV RNA (based on an assay considered sensitive at the time of treatment) at the end of treatment with a pegylated interferon-based regimen, but HCV RNA detectable within 24 weeks of treatment follow up
4. HCV RNA =1,000 IU/mL at screening
5. Documentation of a liver biopsy within 3 years or fibroscan within 6 months prior to randomisation
6. Age 18 to 70 years
7. Female patients:

   1. with documented hysterectomy,
   2. who have had both ovaries removed,
   3. with documented tubal ligation,
   4. who are post-menopausal with last menstrual period at least 12 months prior to screening, or
   5. of childbearing potential with a negative serum pregnancy test at screening and Day 1, that, if sexually active, agree to use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin in addition to the consistent and correct use of a condom. Patients must agree not to breast-feed at any time from the date of screening until 7 months after the last dose of ribavirin
   6. Medically accepted methods of contraception for females in this trial are ethinyl estradiol-containing contraceptives, diaphragm with spermicide substance, and intra uterine device.

   Male patients:
   1. who are documented to be sterile, or
   2. who are without pregnant female partner(s) and consistently and correctly use a condom while their female partner(s) (if of child-bearing potential) use one of the appropriate medically accepted methods of birth control from the date of screening until 7 months after the last dose of ribavirin. It is in the responsibility of the male patient to ensure that his partner(s) is not pregnant prior to screening into the study or becomes pregnant during the treatment and the observation phase. Female partners of childbearing potential should perform monthly pregnancy tests from the date of screening until 7 months after the last dose of ribavirin (tests will be provided by the sponsor)
8. Signed informed consent form prior to trial participation

Exclusion criteria:

1. HCV infection of mixed genotype (1/2, 1/3, and 1/4) diagnosed by genotypic testing at screening
2. Evidence of acute or chronic liver disease due to causes other than chronic HCV infection. Incidental steatosis diagnosed by biopsy is not an exclusion criterion
3. HIV co-infection
4. Hepatitis B virus (HBV) infection based on presence of hepatitis B surface Antigen (HBs-Ag)
5. Active malignancy, or history of malignancy within the last 5 years prior to screening (with an exception of appropriately treated basal cell carcinoma of the skin or in situ carcinoma of the uterine cervix)
6. Active or, history of alcohol or illicit drug abuse other than cannabis within the past 12 months
7. A condition that is defined as one which in the opinion of investigator may put the patient at risk because of participation in this study, may influence the results of this study, or limit the patient's ability to participate in this study
8. Usage of any investigational drugs within 30 days prior to screening, or planned usage of an investigational drug during the course of this study
9. Received concomitant systemic antiviral, hematopoietic growth factor, or immunomodulatory treatment within 30 days prior to randomisation.Patients being treated with oral antivirals such as acyclovir, famciclovir or valacyclovir for recurrent herpes simplex infection; or with oseltamivir or zanamivir for influenza A infection, may be screened
10. Received silymarin (milk thistle), glycyrrhizin, or Sho-saiko-to (SST) within 28 days prior to randomisation and throughout the treatment phase
11. Patients who have been previously treated with at least one dose of any antiviral or immunomodulatory drug other than interferon alfa or ribavirin for acute or chronic HCV infection including and not restricted to protease or polymerase inhibitors
12. Known hypersensitivity to any ingredient of the study drugs
13. Alpha fetoprotein value >100 ng/mL at screening; if >20 ng/mL and =100 ng/mL, patients may be included if there is no evidence of liver cancer in an appropriate imaging study (e.g., ultrasound, computed tomography (CT) scan, or magnetic resonance imaging (MRI)) within last 6 months prior to randomisation (Visit 2) Other exclusion criteria related to pegylated interferon-a and/or ribavirin restrictions are not listed here.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-09; Primary Completion 2015-10 (Estimated)

PRIMARY OUTCOMES:
Sustained Virological Response 12 weeks post-treatment (SVR12): Plasma Hepatitis C Virus (HCV) Ribonucleic Acid ( RNA) <25 IU/mL undetected at 12 weeks after the originally planned treatment duration. | 60 weeks

SECONDARY OUTCOMES:
Virological response after 24 weeks of treatment discontinuation (SVR24): Plasma HCV RNA level <25 IU/mL, undetected; 24 weeks after the originally planned treatment duration | 72 weeks
Early Treatment Success (ETS): Plasma HCV RNA level <25 IU/mL (detected or undetected) at Week 4 and HCV RNA <25 IU/mL, undetected at Week 8 | 8 weeks
Alanine Aminotransferase (ALT) and Aspartate Aminotransferase (AST) normalisation. ALT and AST normal at end of treatment and post treatment. | 72 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim